CLINICAL TRIAL: NCT00126399
Title: A Clinical Trial to Determine the Effects of 40 Mg Doxycycline Versus a Placebo Control for the Treatment of Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CollaGenex Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COL-101-ROSE-301+302
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Last update posted 2005-08-19 (Estimated); Status verified 2005-08

CONDITIONS: Rosacea
Keywords: rosacea; acne rosacea
MeSH Terms: conditions — Rosacea | interventions — Doxycycline

INTERVENTIONS:
Drug: doxycycline

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of 40 mg doxycycline controlled-release capsules administered once daily for the treatment of rosacea compared with a placebo.

ELIGIBILITY:
Main Inclusion Criteria:

* Healthy patients with rosacea
* Males and females ≥18 years of age
* 10 to 40 papules and pustules and ≤2 nodules
* Score of 2 to 4 on the IGA
* Presence of telangiectasia
* Moderate to severe erythema

Main Exclusion Criteria:

* Use of topical acne treatments or topical or systemic antibiotics
* Use of systemic retinoids within 90 days of baseline
* Use of an investigational drug within 90 days of baseline
* Pregnant or nursing women
* Women of childbearing potential not using an adequate form of contraception
* Change in method of contraception within 4 months of baseline
* Known hypersensitivity to tetracyclines
* Surgeries that bypass or exclude the duodenum or achlorhydria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528
Dates: Start 2004-06; Study Completion 2005-04

PRIMARY OUTCOMES:
Change in total inflammatory lesion count

SECONDARY OUTCOMES:
Change from baseline in erythema scale scores
change from baseline in the investigator's global assessment (IGA) score
proportion of patients being clear or near-clear at endpoint